CLINICAL TRIAL: NCT03598790
Title: A Multicenter, Open-Label Study to Assess the Long-Term Safety, Tolerability, and Efficacy of Bimekizumab in Adult Subjects With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: A Study to Evaluate the Efficacy and Safety of Bimekizumab in Adult Subjects With Moderate to Severe Chronic Plaque Psoriasis
Acronym: BE BRIGHT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PS0014; 2016-003427-30 (EudraCT Number)
Record Dates: First submitted 2018-07-16; First posted 2018-07-26 (Actual); Results first posted 2024-12-06 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Chronic Plaque Psoriasis; Moderate to Severe Chronic Plaque Psoriasis
Keywords: Bimekizumab; PSO; Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — bimekizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bimekizumab dose regimen 1 (Experimental): Subjects are randomized to receive either dose regimen 1 (BKZ 1) or dose regimen 2 (BKZ 2) during the 144-week Treatment Period (open-label), those on BKZ 1 will switch to BKZ 2 at Week 24 or later (at the next scheduled clinic visit after Week 48)
  Eligible subjects who completed the Treatment Period (open-label), and have entered Safety Follow Up (SFU) or completed SFU would start OLE2 on BKZ 1 before switching to BKZ 2 after 16 weeks.
  Intervention Name: Bimekizumab
  Interventions: Drug: Bimekizumab
- Bimekizumab dose regimen 2 (Experimental): Subjects are randomized to receive BKZ 2 during the 144-week Treatment Period (open-label).
  Eligible subjects who completed the Treatment Period (open-label), would continue OLE2 on BKZ 2.
  Intervention Name: Bimekizumab
  Interventions: Drug: Bimekizumab

INTERVENTIONS:
Drug: Bimekizumab — Subjects will receive bimekizumab at pre-specified time-points.
  Other Names: UCB4940

SUMMARY:
This is a study to evaluate the long-term safety and tolerability of bimekizumab in adult subjects with moderate to severe chronic plaque psoriasis (PSO).

DETAILED DESCRIPTION:
The study consists of a 144-week Treatment Period (open-label) and an optional 48-week Open-Label Extension Period 2 (OLE2) for eligible subjects in the USA and Canada.

ELIGIBILITY:
Inclusion Criteria:

Treatment Period (open-label)

* Subject is considered reliable and capable of adhering to the protocol (eg, able to understand and complete diaries), visit schedule, and medication intake according to the judgment of the Investigator
* Subject completes the feeder study (PS0008 [NCT03412747], PS0009 [NCT03370133], PS0013 [NCT03410992]) without meeting any withdrawal criteria
* Female subjects must be:

  1. Postmenopausal: Menopause is defined as 12 consecutive months of amenorrhea, for which there is no other obvious pathological or physiological cause
  2. Permanently sterilized (eg, tubal occlusion, hysterectomy, bilateral salpingectomy)
  3. Or, if of childbearing potential (and engaged in sexual activity that could result in procreation), must be willing to use a highly effective method of contraception throughout the duration of the study until 20 weeks after last administration of investigational medicinal product (IMP), and have a negative pregnancy test at the feeder study in final visit/Baseline visit in PS0014

OLE2 Period (USA and Canada)

* Completed the OLE Period without meeting any withdrawal criteria
* Compliant with ongoing clinical study requirements
* Female subject of childbearing potential must be willing to use highly effective method of contraception
* Subjects with a diagnosis of Crohn's disease or ulcerative colitis are allowed as long as they have no active symptomatic disease (US only)
* Signed a separate OLE2 Period ICF

Exclusion Criteria:

Treatment Period (open-label)

* Subject has previously participated in this study
* Female subjects who plan to become pregnant during the study or within 20 weeks following last dose of study medication
* Subject has any medical or psychiatric condition that, in the opinion of the Investigator, could jeopardize or would compromise the subject's ability to participate in this study. Note: For any subject with an ongoing Serious Adverse Event (SAE), or a history of serious infections in the feeder study, the Medical Monitor must be consulted prior to the subject's entry into PS0014, although the decision on whether to enroll the subject remains with the Investigator
* Subject has a positive or indeterminate interferon gamma release assay (IGRA) in a feeder study, unless appropriately evaluated and treated
* Subject may not participate in another study of a medicinal product or device under investigation other than the substudy
* Subject has a history of chronic alcohol or drug abuse within 6 months prior to Baseline as assessed by medical history, site interview, and/or results of the specified urine drug screen

OLE2 Period (USA and Canada)

* Subject has developed any medical or psychiatric condition, which, in the Investigator's judgment, would make the subject unsuitable for inclusion in OLE2 Period
* Subject had a positive or indeterminate interferon-gamma release assay (IGRA) in the OLE study to Week 144, unless appropriately evaluated and treated
* Presence of active suicidal ideation or severe depression
* Subject has developed any active malignancy or history of malignancy prior to the OLE2 Screening Visit EXCEPT treated and considered cured cutaneous squamous or basal cell carcinoma, or in situ cervical cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1353 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (189):
- United States (48):
  - Ps0014 957, Glendale, Arizona
  - Ps0014 946, Phoenix, Arizona
  - Ps0014 910, Bakersfield, California
  - Ps0014 927, Los Angeles, California
  - Ps0014 919, San Diego, California
  - Ps0014 955, San Diego, California
  - Ps0014 943, San Luis Obispo, California
  - Ps0014 967, Santa Monica, California
  - Ps0014 934, Washington D.C., District of Columbia
  - Ps0014 909, Boynton Beach, Florida
  - Ps0014 912, Coral Gables, Florida
  - Ps0014 928, Fort Myers, Florida
  - Ps0014 906, Hollywood, Florida
  - Ps0014 907, Miami, Florida
  - Ps0014 903, Ocala, Florida
  - Ps0014 921, Ormond Beach, Florida
  - Ps0014 936, Tampa, Florida
  - Ps0014 941, Alpharetta, Georgia
  - Ps0014 954, Skokie, Illinois
  - Ps0014 911, Plainfield, Indiana
  - Ps0014 900, West Des Moines, Iowa
  - Ps0014 905, Overland Park, Kansas
  - Ps0014 962, Owensboro, Kentucky
  - Ps0014 922, Baton Rouge, Louisiana
  - Ps0014 944, New Orleans, Louisiana
  - Ps0014 940, Beverly, Massachusetts
  - Ps0014 925, Brighton, Massachusetts
  - Ps0014 917, Troy, Michigan
  - Ps0014 915, Clayton, Missouri
  - Ps0014 958, Omaha, Nebraska
  - Ps0014 901, Portsmouth, New Hampshire
  - Ps0014 908, East Windsor, New Jersey
  - Ps0014 956, Verona, New Jersey
  - Ps0014 947, Buffalo, New York
  - Ps0014 965, Kew Gardens, New York
  - Ps0014 913, New York, New York
  - Ps0014 963, Rochester, New York
  - Ps0014 961, Rocky Mount, North Carolina
  - Ps0014 932, Oklahoma City, Oklahoma
  - Ps0014 920, Portland, Oregon
  - Ps0014 929, Portland, Oregon
  - Ps0014 937, Johnston, Rhode Island
  - Ps0014 945, Greer, South Carolina
  - Ps0014 931, Dallas, Texas
  - Ps0014 924, Houston, Texas
  - Ps0014 914, San Antonio, Texas
  - Ps0014 951, Webster, Texas
  - Ps0014 933, Murray, Utah
- Australia (9):
  - PS0014 7, Campbelltown
  - PS0014 3, Carlton
  - PS0014 8, East Melbourne
  - PS0014 4, Fremantle
  - Ps0014 10, Kogarah
  - PS0014 6, Kogarah
  - PS0014 5, Phillip
  - PS0014 2, Westmead
  - PS0014 9, Woolloongabba
- Belgium (3):
  - Ps0014 50, Brussels
  - Ps0014 51, Charleroi
  - Ps0014 52, Liège
- Canada (23):
  - Ps0014 658, Ajax
  - Ps0014 659, Calgary
  - Ps0014 672, Edmonton
  - Ps0014 673, Halifax
  - Ps0014 671, Hamilton
  - Ps0014 675, Markham
  - Ps0014 663, Mississauga
  - Ps0014 660, Montreal
  - Ps0014 668, North Bay
  - Ps0014 652, Oakville
  - Ps0014 667, Ottawa
  - Ps0014 661, Peterborough
  - Ps0014 665, Québec
  - Ps0014 651, Richmond Hill
  - Ps0014 650, Surrey
  - Ps0014 676, Surrey
  - Ps0014 653, Toronto
  - Ps0014 662, Toronto
  - Ps0014 664, Toronto
  - Ps0014 657, Waterloo
  - Ps0014 669, Windsor
  - Ps0014 670, Windsor
  - Ps0014 674, Winnipeg
- Germany (18):
  - Ps0014 207, Berlin
  - Ps0014 218, Bonn
  - Ps0014 209, Darmstadt
  - Ps0014 203, Dresden
  - Ps0014 214, Erlangen
  - Ps0014 208, Frankfurt
  - Ps0014 210, Friedrichshafen
  - Ps0014 202, Hamburg
  - Ps0014 211, Hamburg
  - Ps0014 220, Hamburg
  - Ps0014 212, Heidelberg
  - Ps0014 215, Lübeck
  - Ps0014 213, Mahlow
  - Ps0014 219, Münster
  - Ps0014 205, Osnabrück
  - Ps0014 217, Schweinfurt
  - Ps0014 200, Schwerin
  - Ps0014 204, Witten
- Hungary (12):
  - Ps0014 252, Budapest
  - Ps0014 254, Budapest
  - Ps0014 255, Budapest
  - Ps0014 261, Budapest
  - Ps0014 256, Debrecen
  - Ps0014 262, Encs
  - Ps0014 251, Gyula
  - Ps0014 253, Orosháza
  - Ps0014 260, Szeged
  - Ps0014 259, Szekszárd
  - Ps0014 250, Szolnok
  - Ps0014 258, Veszprém
- Italy (2):
  - Ps0014 300, Roma
  - Ps0014 303, Roma
- Japan (30):
  - Ps0014 629, Asahikawa
  - Ps0014 605, Bunkyō City
  - Ps0014 607, Chiyoda-ku
  - Ps0014 610, Chūōku
  - Ps0014 601, Fukuoka
  - Ps0014 619, Gifu
  - Ps0014 620, Hamamatsu
  - Ps0014 608, Itabashi-ku
  - Ps0014 609, Kobe
  - Ps0014 600, Kurume
  - Ps0014 622, Matsumoto
  - Ps0014 604, Minatoku
  - Ps0014 623, Morioka
  - Ps0014 621, Nagoya
  - Ps0014 625, Nankoku
  - Ps0014 624, Obihiro
  - Ps0014 611, Osaka
  - Ps0014 614, Osaka
  - Ps0014 603, Sapporo
  - Ps0014 617, Sendai
  - Ps0014 613, Shimotsuke
  - Ps0014 602, Shinagawa-ku
  - Ps0014 612, Shinjuku-ku
  - Ps0014 618, Shinjuku-ku
  - Ps0014 626, Shinjuku-ku
  - Ps0014 628, Shinjuku-ku
  - Ps0014 606, Takaoka
  - Ps0014 615, Tokyo
  - Ps0014 627, Tokyo
  - Ps0014 616, Tsu
- Poland (25):
  - Ps0014 355, Bialystok
  - Ps0014 361, Bialystok
  - Ps0014 362, Bialystok
  - Ps0014 369, Bialystok
  - Ps0014 371, Bydgoszcz
  - Ps0014 352, Gdansk
  - Ps0014 358, Katowice
  - Ps0014 359, Katowice
  - Ps0014 366, Katowice
  - Ps0014 357, Kielce
  - Ps0014 363, Krakow
  - Ps0014 360, Lodz
  - Ps0014 372, Lodz
  - Ps0014 356, Lublin
  - Ps0014 364, Nowa Sól
  - Ps0014 374, Poznan
  - Ps0014 353, Szczecin
  - Ps0014 350, Warsaw
  - Ps0014 351, Warsaw
  - Ps0014 354, Warsaw
  - Ps0014 365, Wroclaw
  - Ps0014 367, Wroclaw
  - Ps0014 368, Wroclaw
  - Ps0014 370, Wroclaw
  - Ps0014 373, Wroclaw
- Russia (7):
  - Ps0014 400, Moscow
  - Ps0014 402, Moscow
  - Ps0014 403, Moscow
  - Ps0014 404, Saint Petersburg
  - Ps0014 405, Saint Petersburg
  - Ps0014 401, Saratov
  - Ps0014 406, Yaroslavl
- South Korea (5):
  - Ps0014 701, Busan
  - Ps0014 702, Gwangju
  - Ps0014 705, Seongnam-si
  - Ps0014 700, Seoul
  - Ps0014 703, Seoul
- Taiwan (2):
  - Ps0014 754, Taipei
  - Ps0014 755, Taipei
- United Kingdom (5):
  - Ps0014 551, Dundee
  - Ps0014 552, Liverpool
  - Ps0014 550, Manchester
  - Ps0014 554, Reading
  - Ps0014 555, Salford

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: http://www.Vivli.org

REFERENCES:
- [Result] Gordon KB, Langley RG, Warren RB, Okubo Y, Stein Gold L, Merola JF, Peterson L, Wixted K, Cross N, Deherder D, Thaci D. Bimekizumab Safety in Patients With Moderate to Severe Plaque Psoriasis: Pooled Results From Phase 2 and Phase 3 Randomized Clinical Trials. JAMA Dermatol. 2022 Jul 1;158(7):735-744. doi: 10.1001/jamadermatol.2022.1185. PMID 35544084
- [Result] Thaci D, Vender R, de Rie MA, Conrad C, Pariser DM, Strober B, Vanvoorden V, Wang M, Madden C, de Cuyper D, Kimball AB. Safety and efficacy of bimekizumab through 2 years in patients with moderate-to-severe plaque psoriasis: longer-term results from the BE SURE randomized controlled trial and the open-label extension from the BE BRIGHT trial. Br J Dermatol. 2023 Jan 23;188(1):22-31. doi: 10.1093/bjd/ljac021. PMID 36689515
- [Result] Gordon KB, Langley RG, Warren RB, Okubo Y, Rosmarin D, Lebwohl M, Peterson L, Madden C, de Cuyper D, Davies O, Thaci D. Bimekizumab safety in patients with moderate-to-severe plaque psoriasis: pooled data from up to 3 years of treatment in randomized phase III trials. Br J Dermatol. 2024 Mar 15;190(4):477-485. doi: 10.1093/bjd/ljad429. PMID 37950894
- [Result] Lebwohl M, Merola JF, Strober B, Armstrong A, Yoshizaki A, Gisondi P, Szilagyi B, Peterson L, de Cuyper D, Cross N, Davies O, Gottlieb AB. Bimekizumab safety in moderate to severe plaque psoriasis: Rates of hepatic events and changes in liver parameters over 2 years in randomized phase 3/3b trials. J Am Acad Dermatol. 2024 Aug;91(2):281-289. doi: 10.1016/j.jaad.2024.03.041. Epub 2024 Apr 6. PMID 38588819
- [Result] Merola JF, Gottlieb AB, Pinter A, Elewski B, Gooderham M, Warren RB, Piaserico S, Wixted K, Cross N, Tilt N, Wiegratz S, Mrowietz U. Bimekizumab Efficacy in High-Impact Areas: Pooled 2-Year Analysis in Scalp, Nail, and Palmoplantar Psoriasis from Phase 3/3b Randomized Controlled Trials. Dermatol Ther (Heidelb). 2024 Dec;14(12):3291-3306. doi: 10.1007/s13555-024-01295-w. Epub 2024 Nov 22. PMID 39578348
- [Result] Okubo Y, Tada Y, Takahashi H, Abe M, Yamanaka K, Tilt N, Cross N, Deherder D, Matano M, Nakagawa H. Efficacy and Safety of Bimekizumab in Japanese Patients with Generalised Pustular Psoriasis and Erythrodermic Psoriasis: 3-Year Results from BE BRIGHT, a Multicentre, Open-Label, Phase 3 Study. Dermatol Ther (Heidelb). 2025 Oct;15(10):2947-2966. doi: 10.1007/s13555-025-01509-9. Epub 2025 Aug 11. PMID 40788331
- [Result] Strober B, Boehncke WH, Krueger JG, Magnolo N, Vender R, Warren RB, Lopez Pinto JM, Kavanagh S, Hoepken B, Gisondi P. Bimekizumab Efficacy in Psoriasis by Subgroups: Post Hoc Analysis of Phase 3/3b Clinical Trials. Dermatol Ther (Heidelb). 2025 Dec;15(12):3633-3650. doi: 10.1007/s13555-025-01557-1. Epub 2025 Oct 8. PMID 41060492
- [Result] Armstrong A, Papp KA, Lebwohl M, Savage LJ, Yamanaka K, Vlase DE, Warham R, Lambert J, Lopez Pinto JM, Wixted K, Thaci D. Bimekizumab Impact on Patient-Reported Outcomes in Plaque Psoriasis: 4-Year Results from BE SURE, BE VIVID, BE READY, and BE BRIGHT. Dermatol Ther (Heidelb). 2025 Dec 8. doi: 10.1007/s13555-025-01595-9. Online ahead of print. PMID 41359217
- [Derived] Merola JF, Warren RB, Thaci D, Gordon KB, Nishida E, Strober B, Conrad C, Kavanagh S, Lopez Pinto JM, Hoepken B, Gisondi P. Bimekizumab Complete Clearance of Both Skin and Nail Psoriasis: Comparative Efficacy in Phase III/IIIb Studies. Am J Clin Dermatol. 2025 Nov;26(6):967-979. doi: 10.1007/s40257-025-00968-2. Epub 2025 Aug 31. PMID 40886218
- [Derived] Kokolakis G, Warren RB, Strober B, Blauvelt A, Puig L, Morita A, Gooderham M, Korber A, Vanvoorden V, Wang M, de Cuyper D, Madden C, Nunez Gomez N, Lebwohl M. Bimekizumab efficacy and safety in patients with moderate-to-severe plaque psoriasis who switched from adalimumab, ustekinumab or secukinumab: results from phase III/IIIb trials. Br J Dermatol. 2023 Feb 22;188(3):330-340. doi: 10.1093/bjd/ljac089. PMID 36751950

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in September 2018 and concluded in November 2023. Participant flow refers to the Cohort A Safety Set, Cohort A OLE2 Period Set and Cohort B Safety Set. Participants who enrolled in PS0014 after completion of Phase 3 feeder studies were included in Cohort A. An additional Cohort B was added in Japan.
Pre-assignment Details: Cohort A has Treatment Period (TP) (144 wks) followed by SFU Visit (20 wks after final dose). Cohort B has Screening Period (2 to 5 wks) and TP (144 wks) followed by SFU Visit (20 wks after final dose). After Protocol Amendment 3.3 (US) and 3.4 (Canada), 48-week OLE2 Period followed by SFU2 Visit (20 wks after final dose) was added in Cohort A.
Groups:
- Cohort A: BKZ 320 mg Q8W: Based on the PASI90 response and the treatment/dose the participant was receiving in the feeder studies (PS0008 [NCT03412747], PS0009 [NCT03370133], and PS0013 [NCT03410992]), participants were randomized to receive BKZ 320 milligrams (mg) subcutaneously (sc) every 8 weeks (Q8W) in this study during the 144-week (wk) Treatment Period. The BKZ 320 mg Q8W group consisted of all participants who received only Q8W during PS0014 study and did not switch dosing regimen at any time point.
- Cohort A: BKZ 320 mg Q4W/Q8W: Based on the PASI90 response and the treatment/dose the participant was receiving in the feeder study, participants were randomized to receive BKZ 320 mg sc every 4 weeks (Q4W) in this study during the 144-week Treatment Period. The participants switched to BKZ 320 mg Q8W as per protocol. The BKZ 320mg Q4W/Q8W group consisted of all participants who switched from Q4W to Q8W dosing at any of the scheduled switching time points during the study.
- Cohort A: BKZ 320 mg Q4W: Based on the PASI90 response and the treatment/dose the participant was receiving in the feeder study, participants were randomized to receive BKZ 320 mg sc Q4W in this study during the 144-week Treatment Period. The BKZ 320 mg Q4W group consisted of participants who discontinued prior to the planned change of dosing interval from BKZ 320 mg Q4W to BKZ 320 mg Q8W.
- Cohort A: Group A BKZ 320 mg Q8W: Participants who completed the Treatment Period (Week 0 to Week 144) were directly rolled over to the Open-Label Extension 2 (OLE2) Period. Participants continued receiving BKZ 320 mg sc Q8W for 40 additional weeks (from Week 144/OLE2 Period Baseline Visit to OLE2 Period Week 48).
- Cohort A: Group B BKZ 320 mg Q8W: Participants who had completed the Treatment Period Week 144 Visit and who were in the SFU or had completed the SFU at the time of Protocol Amendment 3.3 and 3.4 implementation reinitiated BKZ treatment in the OLE2 Period after 4-week OLE2 Screening Period. Participants in OLE2 Period Group B with an IGA score <3 upon entry received BKZ 320 mg sc Q8W from the Week 144/OLE2 Period Baseline Visit to OLE2 Period Week 48.
- Cohort A: Group B BKZ 320 mg Q4W/Q8W: Participants who had completed the Treatment Period Week 144 Visit and who were in the Safety Follow-Up (SFU) or had completed the SFU at the time of Protocol Amendment 3.3 and 3.4 implementation reinitiated BKZ treatment in the OLE2 Period after 4-week OLE2 Screening Period. Participants with an Investigator's Global Assessment (IGA) score greater than equal to (>=) 3 upon entry in the OLE2 Period received BKZ 320 mg sc Q4W for the first 16 weeks, and then switched to BKZ 320 mg Q8W until OLE2 Period Week 48.
- Cohort B: PSO BKZ Total: Participants with chronic plaque psoriasis (PSO) in Cohort B received BKZ 320 mg sc Q4W until Week 16 and 320 mg Q8W thereafter through Week 40. At Week 48, Cohort B participants with chronic plaque PSO continued BKZ 320 mg Q8W up to Week 144. If the participant's dosing interval had changed to BKZ 320 mg Q4W under Protocol Amendment 1.2, the participant's dosing interval changed to BKZ 320 mg Q8W at the next scheduled clinic visit after implementation of Protocol Amendment 3.2.
- Cohort B: EP BKZ Total: Participants with erythrodermic psoriasis (EP) in Cohort B received BKZ 320 mg sc Q4W until Week 16. Based on IGA response, participants received either BKZ 320 mg sc Q4W or BKZ 320 mg sc Q8W up to Week 144.
- Cohort B: GPP BKZ Total: Participants with generalized pustular psoriasis (GPP) in Cohort B received BKZ 320 mg sc Q4W until Week 16. Based on IGA response, participants received either BKZ 320 mg sc Q4W or BKZ 320 mg sc Q8W up to Week 144.
Period: Treatment Period (TP): Wk0-Wk144
Arm/Group | Cohort A: BKZ 320 mg Q8W | Cohort A: BKZ 320 mg Q4W/Q8W | Cohort A: BKZ 320 mg Q4W | Cohort A: Group A BKZ 320 mg Q8W | Cohort A: Group B BKZ 320 mg Q8W | Cohort A: Group B BKZ 320 mg Q4W/Q8W | Cohort B: PSO BKZ Total | Cohort B: EP BKZ Total | Cohort B: GPP BKZ Total
Started | 384 | 833 | 70 | 0 | 0 | 0 | 45 | 11 | 10
Completed | 326 | 746 | 0 | 0 | 0 | 0 | 38 | 10 | 8
Not Completed | 58 | 87 | 70 | 0 | 0 | 0 | 7 | 1 | 2
Not completed — Adverse Event | 24 | 33 | 24 | 0 | 0 | 0 | 3 | 1 | 2
Not completed — Lack of Efficacy | 4 | 7 | 5 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Protocol Violation | 1 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 7 | 11 | 14 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Consent withdrawn by subject | 14 | 26 | 17 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Covid-19 Pandemic Circumstances | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Long IP pause; Investigator decided termination | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawn By Sponsor | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Patient Did Not Comply With Safety Precautions | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Covid-19 Pandemic Circumstances | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor's Decision | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Unplanned Elective Surgery | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Non-Compliance | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Site Closure; Subject did not want to transfer | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — COVID-19 restrictions; Subject unable to return | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Subject Withdraw Consent (Fear Of Another Ae) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — The Subject Can't Visit the Hospital Anymore | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Completed treatment but missed Week 144 visit | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Non-Compliance-PI early terminated the subject | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: OLE2 Period: Wk 144/OLE2 BL- OLE2 Wk 48
Arm/Group | Cohort A: BKZ 320 mg Q8W | Cohort A: BKZ 320 mg Q4W/Q8W | Cohort A: BKZ 320 mg Q4W | Cohort A: Group A BKZ 320 mg Q8W | Cohort A: Group B BKZ 320 mg Q8W | Cohort A: Group B BKZ 320 mg Q4W/Q8W | Cohort B: PSO BKZ Total | Cohort B: EP BKZ Total | Cohort B: GPP BKZ Total
Started | 0 | 0 | 0 | 226 | 51 | 41 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 216 | 49 | 39 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 10 | 2 | 2 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0
Not completed — Consent withdrawn | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Pt Cannot Commit To Study Schedule | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Cohort A Safety Set (CA-SS) which consisted of all Cohort A study participants who received at least 1 dose of the investigational medicinal product (IMP) in this study and Cohort B Safety Set (CB-SS) which consisted of all Cohort B study participants in the Cohort B Enrolled Set (CB-ES) who received at least 1 dose of IMP in PS0014 study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: BKZ 320 mg Q8W | Cohort A: BKZ 320 mg Q4W/Q8W | Cohort A: BKZ 320 mg Q4W | Cohort B: PSO BKZ Total | Cohort B: EP BKZ Total | Cohort B: GPP BKZ Total | Total
Number analyzed (Participants) | 384 | 833 | 70 | 45 | 11 | 10 | 1353
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (13.7) | 45.5 (13.2) | 45.4 (13.4) | 48.8 (11.5) | 55.3 (11.9) | 46.0 (12.5) | 45.6 (13.3)
Age, Customized [Count of Participants; unit: Participants]
  18 - <65 years | 349 | 757 | 68 | 42 | 10 | 10 | 1236
  65 - <85 years | 35 | 76 | 2 | 3 | 1 | 0 | 117
  >= 85 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 221 | 24 | 9 | 0 | 4 | 376
  Male | 266 | 612 | 46 | 36 | 11 | 6 | 977
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaskan Native | 1 | 1 | 0 | 0 | 0 | 0 | 2
  Asian | 31 | 107 | 8 | 45 | 11 | 10 | 212
  Black | 1 | 14 | 2 | 0 | 0 | 0 | 17
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 0 | 0 | 0 | 0 | 4
  White | 344 | 695 | 58 | 0 | 0 | 0 | 1097
  Other/mixed | 5 | 14 | 2 | 0 | 0 | 0 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 40 | 11 | 0 | 0 | 0 | 71
  Not Hispanic or Latino | 364 | 793 | 59 | 45 | 11 | 10 | 1282

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment Emergent Adverse Events (TEAEs) Adjusted by Duration of Subject Exposure to Investigational Medicinal Product (IMP)
Description: The number of TEAEs adjusted by duration of exposure to study treatment were scaled such that it provides an incidence rate per 100 patient-years. If a participant had multiple events, the time of exposure was calculated to first occurrence of the AE being considered. If a participant had no events, the total time at risk was used.
Time Frame: From Baseline up to 165 weeks for each study participant not entering the OLE2 Period and up to 212 weeks for participants entering OLE2 Period
Population: CA-SS -All Cohort A participants who received at least 1 dose of the IMP in this study. Cohort A OLE2 Period Set (CA-OL2S)-All participants who received at least 1 dose of BKZ in the OLE2 Period. Cohort B PSO SS-All participants with a diagnosis of PSO disease at Baseline. Cohort B EP-SS-All participants with a diagnosis of EP disease at Baseline. Cohort B GPP-SS-All participants with a diagnosis of GPP disease at Baseline.
Measure: Number (95% Confidence Interval); unit: no. of new events per 100 subject-years
Groups:
- Cohort A: BKZ 320 mg Q8W: Participants who received BKZ 320 mg Q8W and who switched from Q4W to Q8W dosing at any of the scheduled time points during the 144-week Treatment Period. The participants who switched from BKZ 320 mg Q4W to Q8W during the study were included in both the BKZ 320 mg Q4W group and the BKZ 320 mg Q8W group.
- Cohort A: BKZ 320 mg Q4W: Participants who received BKZ 320 mg Q4W during the 144-week Treatment Period. The participants who switched from BKZ 320 mg Q4W to Q8W during the study were included in both the BKZ 320 mg Q4W group and the BKZ 320 mg Q8W group.
Arm/Group | Cohort A: BKZ 320 mg Q8W | Cohort A: BKZ 320 mg Q4W | Cohort A: Group A BKZ 320 mg Q8W | Cohort A: Group B BKZ 320 mg Q8W | Cohort A: Group B BKZ 320 mg Q4W/Q8W | Cohort B: PSO BKZ Total | Cohort B: EP BKZ Total | Cohort B: GPP BKZ Total
Number analyzed (Participants) | 1217 | 903 | 226 | 51 | 41 | 45 | 11 | 10
no. of new events per 100 subject-years | 97.83 [91.73 to 104.22] | 179.68 [166.62 to 193.49] | 79.02 [65.97 to 93.89] | 77.11 [51.64 to 110.74] | 73.78 [47.75 to 108.92] | 244.08 [178.03 to 326.60] | 328.25 [163.86 to 587.33] | 188.71 [86.29 to 358.22]

2. Secondary Outcome: Number of Serious Adverse Events (SAEs) Adjusted by Duration of Subject Exposure to IMP
Description: The number of SAEs adjusted by duration of exposure to study treatment were scaled such that it provides an incidence rate per 100 patient-years. If a participant had multiple events, the time of exposure was calculated to the first occurrence of the AE being considered. If a participant had no events, the total time at risk is used.
Time Frame: as for outcome 1
Population: CA-SS -All Cohort A participants who received at least 1 dose of the IMP in this study. CA-OL2S-All participants who received at least 1 dose of BKZ in the OLE2 Period. Cohort B PSO SS-All participants with a diagnosis of PSO disease at Baseline. Cohort B EP-SS-All participants with a diagnosis of EP disease at Baseline. Cohort B GPP-SS-All participants with a diagnosis of GPP disease at Baseline.
Measure: Number (95% Confidence Interval); unit: no. of new events per 100 subject-years
Arm/Group | Cohort A: BKZ 320 mg Q8W | Cohort A: BKZ 320 mg Q4W | Cohort A: Group A BKZ 320 mg Q8W | Cohort A: Group B BKZ 320 mg Q8W | Cohort A: Group B BKZ 320 mg Q4W/Q8W | Cohort B: PSO BKZ Total | Cohort B: EP BKZ Total | Cohort B: GPP BKZ Total
Number analyzed (Participants) | 1217 | 903 | 226 | 51 | 41 | 45 | 11 | 10
no. of new events per 100 subject-years | 5.24 [4.36 to 6.25] | 6.72 [5.19 to 8.56] | 4.44 [2.22 to 7.95] | 9.05 [2.94 to 21.13] | 8.93 [2.43 to 22.86] | 5.86 [2.36 to 12.08] | 19.51 [6.34 to 45.54] | 7.56 [0.92 to 27.32]

3. Secondary Outcome: Number of TEAEs Leading to Withdrawal Adjusted by Duration of Subject Exposure to IMP
Description: The number of TEAEs leading to withdrawal adjusted by duration of exposure to study treatment were scaled such that it provided an incidence rate per 100 patient-years. If a participant had multiple events, the time of exposure was calculated to the first occurrence of the AE being considered. If a participant had no events, the total time at risk was used.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: no. of new events per 100 subject-years
Arm/Group | Cohort A: BKZ 320 mg Q8W | Cohort A: BKZ 320 mg Q4W | Cohort A: Group A BKZ 320 mg Q8W | Cohort A: Group B BKZ 320 mg Q8W | Cohort A: Group B BKZ 320 mg Q4W/Q8W | Cohort B: PSO BKZ Total | Cohort B: EP BKZ Total | Cohort B: GPP BKZ Total
Number analyzed (Participants) | 1217 | 903 | 226 | 51 | 41 | 45 | 11 | 10
no. of new events per 100 subject-years | 2.11 [1.57 to 2.76] | 2.59 [1.69 to 3.80] | 0.79 [0.10 to 2.86] | 1.77 [0.04 to 9.86] | 4.37 [0.53 to 15.79] | 2.42 [0.50 to 7.08] | 3.27 [0.08 to 18.19] | 7.68 [0.93 to 27.74]

4. Secondary Outcome: Psoriasis Area Severity Index 90 (PASI90) Response at Week 144 (Non-responder Imputation)
Description: The PASI90 response assessments were based on improvement (reduction) of at least 90% in the PASI score compared to Baseline. Body divided into 4 areas: head, arms, trunk to groin, and legs to top of buttocks. Assignment of an average score for redness, thickness, and scaling for each of the 4 body areas with score of 0 (clear) to 4 (very marked). Determining the percentage of skin covered with PSO for each of the body areas and converting to a 0 to 6 scale. Final PASI=average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of the respective section, and weighted by the percentage of the person's affected skin for respective section. The minimum possible PASI score is 0= no disease, the maximum score is 72= maximal disease.
Time Frame: Week 144 compared to Baseline of Feeder study for Cohort A and Baseline of PS0014 for Cohort B
Population: Cohort A FAS included all Cohort A enrolled study participants who received at least 1 dose of IMP and had a valid efficacy measurement for PASI at Baseline of the feeder study and at Baseline of this study. Cohort B Psoriasis FAS included study participants with chronic plaque PSO at Baseline. Study participants who had missing data at the Week 144 were treated as though they did not respond to the treatment using Non-responder imputation (NRI) method.
Measure: Number; unit: percentage of participants
Groups:
- Cohort A: BKZ 320mg Q4W: Based on the PASI90 response and the treatment/dose the participant was receiving in the feeder study, participants were randomized to receive BKZ 320 mg sc Q4W in this study during the 144-week Treatment Period. The BKZ 320 mg Q4W group consisted of participants who discontinued prior to the planned change of dosing interval from BKZ 320 mg Q4W to BKZ 320 mg Q8W.
Arm/Group | Cohort A: BKZ 320 mg Q8W | Cohort A: BKZ 320 mg Q4W/Q8W | Cohort A: BKZ 320mg Q4W | Cohort B: PSO BKZ Total
Number analyzed (Participants) | 384 | 832 | 70 | 45
percentage of participants | 77.6 | 80.2 | 0 | 73.3

5. Secondary Outcome: Psoriasis Area Severity Index 90 (PASI90) Response at Week 144 (Observed Case)
Description: PASI90 response assessments were based on improvement (reduction) of at least 90% in the PASI score compared to Baseline. Body divided into 4 areas: head, arms, trunk to groin, and legs to top of buttocks. Assignment of an average score for redness, thickness, and scaling for each of the 4 body areas with score of 0 (clear) to 4 (very marked). Determining the percentage of skin covered with PSO for each of the body areas and converting to a 0 to 6 scale. Final PASI=average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by involved psoriasis area score of respective section, and weighted by percentage of person's affected skin for respective section. Minimum score is 0= no disease, maximum score is 72= maximal disease.
Time Frame: Week 144 compared to Baseline of PS0014 for Cohort B
Population: Cohort B GPP FAS included study participants with GPP at Baseline. Cohort B EP FAS included study participants with EP at Baseline. Only study participants with available data who had not discontinued study treatment at Week 144 were considered for the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort B: EP BKZ Total | Cohort B: GPP BKZ Total
Number analyzed (Participants) | 11 | 10
percentage of participants | 90.0 | 85.7

6. Secondary Outcome: Investigator´s Global Assessment (IGA) 0/1 Response at Week 144 (Non-responder Imputation)
Description: The Investigator assessed the overall severity of psoriasis using the following 5-point scale: 0 = Clear (no signs of psoriasis; post-inflammatory hyperpigmentation may be present); 1= Almost clear (no thickening; normal to pink coloration; no to minimal focal scaling); 2= Mild (just detectable to mild thickening; pink to light red coloration; predominately fine scaling); 3= Moderate (clearly distinguishable to moderate thickening; dull to bright red coloration; moderate scaling); 4= Severe (Severe thickening with hard edges; bright to deep dark red coloration; severe/coarse scaling covering almost all or all lesions). IGA response -IGA score of clear [0] or almost clear [1] with at least two category improvement from Baseline at visit timepoint.
Time Frame: Week 144 compared to Baseline of Feeder study for Cohort A and Baseline of PS0014 for Cohort B
Population: Cohort A FAS included all Cohort A enrolled study participants who received at least 1 dose of IMP and had a valid efficacy measurement for PASI at Baseline of the feeder study and at Baseline of this study. Cohort B Psoriasis FAS included study participants with chronic plaque PSO at Baseline. Study participants who had missing data at the Week 144 were treated as though they did not respond to the treatment using NRI.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: BKZ 320 mg Q8W | Cohort A: BKZ 320 mg Q4W/Q8W | Cohort A: BKZ 320 mg Q4W | Cohort B: PSO BKZ Total
Number analyzed (Participants) | 384 | 832 | 70 | 45
percentage of participants | 76.8 | 79.0 | 0 | 60.0

7. Secondary Outcome: Investigator´s Global Assessment (IGA) 0/1 Response at Week 144 (Observed Case)
Description: The Investigator assessed the overall severity of psoriasis using the following 5-point scale: 0 = Clear (no signs of psoriasis; post-inflammatory hyperpigmentation may be present); 1= Almost clear (no thickening; normal to pink coloration; no to minimal focal scaling); 2= Mild (just detectable to mild thickening; pink to light red coloration; predominately fine scaling); 3= Moderate (clearly distinguishable to moderate thickening; dull to bright red coloration; moderate scaling); 4= Severe (Severe thickening with hard edges; bright to deep dark red coloration; severe/coarse scaling covering almost all or all lesions). IGA response -IGA score of 0 or 1 at Week 144.
Time Frame: Week 144 for Cohort B EP and GPP groups
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Cohort B: EP BKZ Total | Cohort B: GPP BKZ Total
Number analyzed (Participants) | 11 | 10
percentage of participants | 80.0 | 85.7

ADVERSE EVENTS:
Time Frame: From Baseline up to 165 weeks for each study participant not entering the OLE2 Period and up to 212 weeks for participants entering OLE2 Period
Description: TEAEs were defined as events that have a start date on or following the first administration of study treatment in PS0014 through the final administration of study treatment + 140 days (covering the 20-week SFU Period). Cohort A OLE2 Period Set (CA-OL2S) included all participants who received at least 1 dose of BKZ in the OLE2 Period. SS was used.
Groups:
- Cohort A: BKZ 320 mg Q8W: Participants who received BKZ 320 mg Q8W and who switched from Q4W to Q8W dosing at any of the scheduled time points during the 144-week Treatment Period. The participants who switched from BKZ 320 mg Q4W to Q8W during the study were included in both the BKZ 320 mg Q4W group and the BKZ 320 mg Q8W group. All the adverse events occurred during the BKZ 320 mg Q8W treatment at any timepoint of the study were included in this arm.
- Cohort A: BKZ 320 mg Q4W: Participants who received BKZ 320 mg Q4W during the 144-week Treatment Period. The participants who switched from BKZ 320 mg Q4W to Q8W during the study were included in both the BKZ 320 mg Q4W group and the BKZ 320 mg Q8W group. All the adverse events occurred during the BKZ 320 mg Q4W treatment at any timepoint of the study were included in this arm.
Arm/Group | Cohort A: BKZ 320 mg Q8W | Cohort A: BKZ 320 mg Q4W | Cohort A: Group A BKZ 320 mg Q8W | Cohort A: Group B BKZ 320 mg Q8W | Cohort A: Group B BKZ 320 mg Q4W/Q8W | Cohort B: PSO BKZ Total | Cohort B: EP BKZ Total | Cohort B: GPP BKZ Total
All-Cause Mortality (participants affected / at risk) | 9/1217 | 6/903 | 0/226 | 0/51 | 0/41 | 0/45 | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 124/1217 | 65/903 | 11/226 | 5/51 | 4/41 | 7/45 | 5/11 | 2/10
Other Adverse Events (participants affected / at risk) | 771/1217 | 566/903 | 97/226 | 16/51 | 21/41 | 43/45 | 11/11 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Cohort A: BKZ 320 mg Q8W (N=1217) | Cohort A: BKZ 320 mg Q4W (N=903) | Cohort A: Group A BKZ 320 mg Q8W (N=226) | Cohort A: Group B BKZ 320 mg Q8W (N=51) | Cohort A: Group B BKZ 320 mg Q4W/Q8W (N=41) | Cohort B: PSO BKZ Total (N=45) | Cohort B: EP BKZ Total (N=11) | Cohort B: GPP BKZ Total (N=10)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wolff-Parkinson-White syndrome (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 3 (3) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperparathyroidism primary (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal prolapse (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0/0 (0) | 0/0 (0)
Oroantral fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stent-graft endoleak (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystocholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bursitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoas abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Streptococcal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corona virus infection (Infections and infestations) | 13 (13) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal column injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inclusion body myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Kyphosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral artery embolism (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemiplegic migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Relapsing-remitting multiple sclerosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intercostal neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spondylitic myelopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pregnancy on oral contraceptive (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bipolar I disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug dependence (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic aneurysm rupture (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femoral artery embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythrodermic psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: BKZ 320 mg Q8W (N=1217) | Cohort A: BKZ 320 mg Q4W (N=903) | Cohort A: Group A BKZ 320 mg Q8W (N=226) | Cohort A: Group B BKZ 320 mg Q8W (N=51) | Cohort A: Group B BKZ 320 mg Q4W/Q8W (N=41) | Cohort B: PSO BKZ Total (N=45) | Cohort B: EP BKZ Total (N=11) | Cohort B: GPP BKZ Total (N=10)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac hypertrophy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 5 (5) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 12 (14) | 6 (6) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 8 (8) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Dry eye (Eye disorders) | 4 (4) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 24 (27) | 19 (20) | 2 (2) | 0 (0) | 0 (0) | 7 (8) | 0 (0) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 14 (15) | 17 (17) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 14 (14) | 7 (7) | 2 (3) | 0 (0) | 1 (1) | 7 (8) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 11 (12) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 11 (13) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 8 (8) | 5 (7) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 6 (6) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 5 (5) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (7) | 1 (1) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Glossitis (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0)
Coating in mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 25 (30) | 8 (9) | 3 (3) | 0 (0) | 0 (0) | 10 (11) | 1 (1) | 3 (4)
Peripheral swelling (General disorders) | 8 (9) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 5 (5) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 10 (10) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 152 (223) | 174 (230) | 14 (15) | 1 (1) | 1 (1) | 19 (25) | 7 (9) | 2 (2)
Oral candidiasis (Infections and infestations) | 127 (238) | 145 (234) | 13 (18) | 3 (5) | 6 (6) | 11 (18) | 4 (4) | 2 (2)
Corona virus infection (Infections and infestations) | 174 (187) | 18 (18) | 34 (35) | 3 (3) | 8 (8) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 97 (127) | 74 (85) | 12 (14) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 58 (79) | 49 (72) | 6 (8) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 24 (30) | 35 (43) | 1 (1) | 1 (1) | 1 (2) | 7 (11) | 1 (2) | 1 (1)
Pharyngitis (Infections and infestations) | 27 (28) | 19 (22) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 20 (22) | 25 (30) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 17 (19) | 13 (15) | 1 (1) | 1 (1) | 1 (3) | 5 (7) | 1 (1) | 1 (2)
Oral herpes (Infections and infestations) | 15 (19) | 16 (18) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 1 (3)
Angular cheilitis (Infections and infestations) | 14 (15) | 14 (18) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 16 (16) | 12 (13) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 12 (13) | 9 (11) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 10 (11) | 7 (8) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Cystitis (Infections and infestations) | 9 (11) | 4 (5) | 2 (2) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Skin bacterial infection (Infections and infestations) | 3 (3) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 3 (4) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 5 (7) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
Tinea cruris (Infections and infestations) | 5 (5) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Genital candidiasis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 10 (10) | 8 (8) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 9 (12) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 7 (7) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 5 (6) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 19 (23) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 15 (17) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 12 (14) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 9 (9) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
White blood cell count decreased (Investigations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 13 (14) | 8 (8) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 11 (11) | 9 (9) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 12 (12) | 6 (6) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 7 (7) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 48 (55) | 19 (22) | 0 (0) | 0 (0) | 1 (1) | 4 (6) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 28 (31) | 23 (24) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 26 (27) | 5 (5) | 5 (5) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 9 (10) | 9 (11) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 5 (7) | 7 (8) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 7 (8) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 7 (10) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 55 (61) | 20 (27) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 27 (30) | 21 (22) | 5 (5) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 16 (16) | 15 (15) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 5 (5) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 44 (52) | 16 (18) | 3 (4) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 34 (38) | 25 (32) | 2 (2) | 2 (2) | 4 (5) | 6 (9) | 0 (0) | 1 (2)
Eczema (Skin and subcutaneous tissue disorders) | 30 (42) | 17 (21) | 1 (1) | 0 (0) | 0 (0) | 15 (28) | 3 (3) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 15 (15) | 10 (11) | 1 (1) | 0 (0) | 1 (1) | 1 (3) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 13 (13) | 6 (7) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 14 (14) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 9 (9) | 9 (9) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 6 (7) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 6 (7) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 6 (7) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0)
Erythrodermic psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Milia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 55 (55) | 33 (34) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-10-12): https://cdn.clinicaltrials.gov/large-docs/90/NCT03598790/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-11): https://cdn.clinicaltrials.gov/large-docs/90/NCT03598790/SAP_001.pdf